CLINICAL TRIAL: NCT01433679
Title: The Effect of a Web-Based Behavioral Intervention on Physical Activity Levels in Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HopeLab Foundation (Other)
Collaborators: West Virginia University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HLZZ-001
Record Dates: First submitted 2011-09-12; First posted 2011-09-14 (Estimated); Last update posted 2012-07-16 (Estimated); Status verified 2012-07

CONDITIONS: Health Behavior; Adolescent Behavior; Motivation
Keywords: Health Behavior; Exercise; Adolescent Behavior; Motivation; Biological Markers
MeSH Terms: conditions — Health Behavior; Adolescent Behavior; Motor Activity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Website intervention (Experimental): Participants randomly assigned to the Website Intervention arm receive access to the motivational rewards website. The website displays the individual's physical activity data and allocates reward points based on the amount and intensity of physical activity. The website also allows reward points to be redeemed for various rewards such as gift cards to retail outlets, donations to charities, small tangible goods, and customization of participants' cartoon-like avatars on the website.
  Interventions: Behavioral: Zamzee Intervention
- Control (No Intervention): Participants in the control group will not have access to the motivational website. No other product or intervention will be introduced to the control group.

INTERVENTIONS:
Behavioral: Zamzee Intervention — The Zamzee intervention is designed to motivate middle school-aged children to increase their rates of moderate to vigorous physical activity (MVPA) by providing rewards based on amount and duration of physical activity. Rewards include gift cards to retail stores, donations to charity, small tangible goods, and customization of their cartoon-like avatars on the website.
  Arms: Website intervention

SUMMARY:
The primary purpose of this study is to test whether rewarding physical activity with a motivational website will increase physical activity levels in middle school-aged children over six months. As a secondary outcome, the study also tests the intervention's impact on biological measures of inflammation and metabolic function in a sub-set of study participants who agree to provide blood samples.

DETAILED DESCRIPTION:
Physical activity is associated with a variety of positive health outcomes, as well as improved metabolic profiles and reduced inflammation. However, levels of moderate to vigorous physical activity (MVPA) diminish dramatically as children move into the middle school years. To address this problem, this study tests a behavioral intervention, called "Zamzee," designed to motivate middle school-aged children to increase their levels of MVPA. The Zamzee intervention consists of a 3-axis accelerometer that tracks individual physical activity rates over time and a website that displays individual physical activity rates and provides rewards for maintaining or improving physical activity rates. The primary aim of this randomized, controlled trial is to test whether middle school-aged children randomly assigned to the Zamzee intervention will show significantly greater levels of physical activity levels over six months, compared with control group participants who wear the accelerometer but have no access to the rewards website. A secondary aim is to test the intervention's impact on biological parameters that may contribute to the long-term health effects of inactivity (including C-reactive protein as a measure of inflammation, and hemoglobin-A1C as a measure of metabolic status) in a sub-set of study participants who agree to provide blood samples.

ELIGIBILITY:
Inclusion Criteria:

* Middle-school-aged students aged 11 to 14

Exclusion Criteria:

* Previously participation in a Zamzee pilot study
* Existing medical conditions or health complications that will interfere with the ability to be physically active
* Inability to read and write English

Ages: 11 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 448 (Actual)
Dates: Start 2011-09; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Physical activity | Six months
  The amount and intensity of physical activity is recorded continuously every study day that participants wear their accelerometer for the duration of the six month study. The primary outcome reported will be rates of "moderate to vigorous physical activity" as defined by the CDC.

SECONDARY OUTCOMES:
Metabolic and inflammatory biomarkers | Six months
  In the subset of study participants who agree to provide blood samples, blood samples collected at study baseline and at the six month study completion will be assayed for measures of inflammation (e.g., C-reactive protein) and metabolic function (e.g.,hemoglobin-A1C).

CONTACTS AND LOCATIONS:
Overall Officials: Jana Haritatos, PhD, Principal Investigator — HopeLab Foundation; Steve Cole, PhD, Study Director — HopeLab Foundation
Locations (6):
- United States (6):
  - Los Osos Middle School, Los Osos, California
  - Berkley Maynard Academy, Oakland, California
  - E.C. Reems Academy, Oakland, California
  - Judkins Middle School, Pismo Beach, California
  - Vista Academy of Visual and Performing Arts, Vista, California
  - West Virginia University, Morgantown, West Virginia